CLINICAL TRIAL: NCT02735980
Title: A Phase 2 Study of LY2606368 in Patients With Extensive Stage Disease Small Cell Lung Cancer
Brief Title: A Study of Prexasertib (LY2606368) in Participants With Extensive Stage Disease Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16015; I4D-MC-JTJH (Other: Eli Lilly and Company); 2015-005069-21 (EudraCT Number)
Record Dates: First submitted 2016-03-31; First posted 2016-04-13 (Estimated); Results first posted 2020-03-17 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2019-05-01

CONDITIONS: Small Cell Lung Cancer
Keywords: SCLC; LY2606368; CHK1
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — prexasertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Prexasertib (Platinum Sensitive Disease) (Experimental): 105 mg/m^2 Intravenous (IV) prexasertib administered of every 14 days with extensive stage disease small cell lung cancer (ED-SCLC) who had platinum-sensitive disease (has prior platinum based therapy with subsequent progression greater or less than 90 days after last dose of platinum based therapy).
  Interventions: Drug: Prexasertib
- Prexasertib (Platinum Resistant Disease) (Experimental): 105 mg/m^2 IV prexasertib administered of every 14 days with extensive stage disease small cell lung cancer (ED-SCLC) who had resistant/refractory disease (did not have an objective response to platinum-based therapy or had progression greater than 90 days after the last dose of platinum).
  Interventions: Drug: Prexasertib
- Prexasertib Exploratory Addendum (Platinum Sensitive Disease) (Experimental): 40 mg/m^2 IV prexasertib Day 1, 2, and Day 3 of a 14 day cycle in participants with ED-SCLC platinum sensitive disease.
  Interventions: Drug: Prexasertib

INTERVENTIONS:
Drug: Prexasertib — Administered IV
  Other Names: LY2606368

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of prexasertib when given to participants with extensive stage disease small cell lung cancer (ED-SCLC). The study will evaluate how the body processes the drug and how the drug affects the body. The study will also evaluate the association between tumor response and the participant's perceived quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Have ED-SCLC and have received a prior platinum-based regimen
* Participants in Cohort 1 and in the addendum must have had an objective response to prior platinum-based therapy with subsequent progression ≥90 days after the last dose of platinum
* Participants in Cohort 2 must have either not had an objective response to prior platinum based therapy or had progression <90 days after the last dose of platinum
* Have a performance status of 0 to 1 on the Eastern Cooperative Oncology Group scale

Exclusion Criteria:

* Have received more than 2 prior therapies for ED-SCLC (including immunotherapy, targeted therapies, or chemotherapy)
* Have symptomatic central nervous system (CNS) malignancy or metastasis. Asymptomatic participants with treated CNS metastases are eligible for this study if they are not currently receiving corticosteroids to treat CNS metastases
* Have previously completed or withdrawn from this study or any other study investigating prexasertib or a checkpoint kinase I (CHK1) inhibitor or have shown hypersensitivity to any of the components of the prexasertib formulation
* Have a serious cardiac condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2016-05-11 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2019-02-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (41):
- United States (14):
  - Highlands Oncology Group, Fayetteville, Arkansas
  - Yale University School of Medicine, New Haven, Connecticut
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Florida Cancer Specialists, Fort Myers, Florida
  - Florida Cancer Specialists and Research Institute, St. Petersburg, Florida
  - Massachusetts General Hospital, Danvers, Massachusetts
  - Washington University Medical Center, St Louis, Missouri
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Chattanooga Oncology Hematology Associates, Chattanooga, Tennessee
  - Sarah Cannon Cancer Center, Nashville, Tennessee
  - Tennessee Oncology PLLC, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - The Center for Cancer and Blood Disorders, Fort Worth, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
- France (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Besançon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lille
  - "For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician.", Montpellier
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vantoux
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Halle, Germany
- Greece (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Athens
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Heraklion
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pátrai
- Netherlands (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Amsterdam
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Breda
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zwolle
- South Korea (2):
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Seoul
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seoul
- Spain (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madrid
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zaragoza
- Turkey (Türkiye) (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Antalya
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Edirne
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Istanbul
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Izmir
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kayseri
- Ukraine (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dnipropetrovsk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kharkiv
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sumy
- United Kingdom (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Headington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leicester
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sheffield

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Jin T, Xu L, Wang P, Hu X, Zhang R, Wu Z, Du W, Kan W, Li K, Wang C, Zhou Y, Li J, Liu T. Discovery and Development of a Potent, Selective, and Orally Bioavailable CHK1 Inhibitor Candidate: 5-((4-((3-Amino-3-methylbutyl)amino)-5-(trifluoromethyl)pyrimidin-2-yl)amino)picolinonitrile. J Med Chem. 2021 Oct 28;64(20):15069-15090. doi: 10.1021/acs.jmedchem.1c00994. Epub 2021 Oct 19. PMID 34665631
- See also: Click here for more information about this study: A Study of Prexasertib (LY2606368) in Participants With Extensive Stage Disease Small Cell Lung Cancer — http://www.lillytrialguide.com/en-US/studies/small-cell%20lung%20cancer/JTJH#?postal=

RESULTS

PARTICIPANT FLOW:
Groups:
- 105 mg/m^2 Prexasertib (Platinum Sensitive Disease): Intravenous (IV) prexasertib (LY2606368)administered on day 1 of every 14 day cycle
- 105 mg/m^2 Prexasertib (Platinum Resistant Disease): IV prexasertib (LY2606368) administered on day 1 of every 14 day cycle
- 40 mg/m2 Prexasertib Exploratory Addendum: 40 mg/m2 IV prexasertib (LY2606368) administered on Days 1, 2 and 3 of a 14-day cycle
Period: Overall Study
Arm/Group | 105 mg/m^2 Prexasertib (Platinum Sensitive Disease) | 105 mg/m^2 Prexasertib (Platinum Resistant Disease) | 40 mg/m2 Prexasertib Exploratory Addendum
Started | 58 | 60 | 15
Received at Least 1 Dose of Study Drug | 56 | 60 | 15
Completed | 48 | 49 | 14
Not Completed | 10 | 11 | 1
Not completed — Adverse Event | 0 | 4 | 1
Not completed — Death | 5 | 4 | 0
Not completed — Physician Decision | 3 | 1 | 0
Not completed — Screen failure | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Prexasertib (Platinum Sensitive Disease): Intravenous (IV) prexasertib (LY2606368)administered on day 1 of every 14 day cycle
- Prexasertib (Platinum Resistant Disease): IV prexasertib (LY2606368) administered on day 1 of every 14 day cycle
- Prexasertib Exploratory Addendum (Platinum Sensitive Disease): IV prexasertib (LY2606368) administered on Days 1, 2 and 3 of a 14-day cycle
- Total: Total of all reporting groups
Arm/Group | Prexasertib (Platinum Sensitive Disease) | Prexasertib (Platinum Resistant Disease) | Prexasertib Exploratory Addendum (Platinum Sensitive Disease) | Total
Number analyzed (Participants) | 58 | 60 | 15 | 133
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.17 (9.21) | 61.45 (7.20) | 61.67 (7.33) | 62.66 (8.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 10 | 4 | 37
  Male | 35 | 50 | 11 | 96
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: N is number of participants with non-missing data.
  Participants
    number analyzed (Participants) | 58 | 59 | 15 | 132
    Hispanic or Latino | 0 | 0 | 0 | 0
    Not Hispanic or Latino | 52 | 53 | 15 | 120
    Unknown or Not Reported | 6 | 6 | 0 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: N is number of participants with non-missing data.
  Participants
    number analyzed (Participants) | 54 | 56 | 15 | 125
    American Indian or Alaska Native | 0 | 0 | 0 | 0
    Asian | 2 | 8 | 2 | 12
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Black or African American | 2 | 1 | 0 | 3
    White | 50 | 47 | 13 | 110
    More than one race | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Greece | 4 | 4 | 0 | 8
  Netherlands | 5 | 1 | 0 | 6
  South Korea | 0 | 8 | 0 | 8
  Turkey | 6 | 15 | 0 | 21
  United States | 24 | 12 | 9 | 45
  Ukraine | 1 | 7 | 0 | 8
  United Kingdom | 2 | 0 | 0 | 2
  France | 7 | 5 | 0 | 12
  Germany | 0 | 2 | 0 | 2
  Spain | 9 | 6 | 6 | 21

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Complete Response (CR) or Partial Response (PR) (Objective Response Rate [ORR])
Description: ORR was the percentage of participants achieving a best overall response (BOR) of complete response (CR) or partial response (PR) as per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. CR defined as the disappearance of all target and non-target lesions and no appearance of new lesions. PR defined as at least a 30% decrease in the sum of the longest diameters (LD) of target lesions (taking as reference the baseline sum LD), no progression of non-target lesions, and no appearance of new lesions
Time Frame: Baseline to 10 months
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Prexasertib (Platinum Sensitive Disease): Intravenous (IV) prexasertib (LY2606368) administered on day 1 of every 14 day cycle
Arm/Group | Prexasertib (Platinum Sensitive Disease) | Prexasertib (Platinum Resistant Disease) | Prexasertib Exploratory Addendum (Platinum Sensitive Disease)
Number analyzed (Participants) | 58 | 60 | 15
percentage of participants | 5.2 [0.7 to 9.6] | 0 [0.0 to 3.7] | 0 [0.0 to 14.8]

2. Secondary Outcome: Pharmacokinetics(PK): Maximum Concentration (Cmax) of Prexasertib Cohort 1 and Cohort 2
Description: Pharmacokinetics(PK): Maximum Concentration of Prexasertib. The same dose was administered to Cohort 1 and Cohort 2 and were combined for analysis.
Time Frame: Cycle 1,3, 5, and 7: Day 1, Day 2 and Day 3- Prior to start of infusion, end of infusion plus 10 minutes, Day 8: anytime
Population: All randomized participants who received at least 1 dose of study drug and had evaluable PK parameters. Cohort 1 and Cohort 2 received the same dose and were combined per protocol.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter
Groups:
- 105 mg/m^2 Prexasertib: IV prexasertib (LY2606368) administered on day 1 of every 14 day cycle
Arm/Group | 105 mg/m^2 Prexasertib
Number analyzed (Participants) | 99
nanogram per milliliter
  Cycle 1 | 722 (64)
  Cycle 3: number analyzed (Participants) | 53
  Cycle 3 | 735 (71)
  Cycle 5: number analyzed (Participants) | 16
  Cycle 5 | 732 (69)
  Cycle 7: number analyzed (Participants) | 5
  Cycle 7 | 1230 (22)

3. Secondary Outcome: Pharmacokinetics(PK): Maximum Concentration of Prexasertib Cohort 3 (40 mg/m^2, Protocol Addenda)
Description: Pharmacokinetics(PK): Maximum Concentration of Prexasertib
Time Frame: as for outcome 2
Population: Al randomized participants with at least 1 dose of study drug, received 40 mg/m^2 and had evaluable PK parameters.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter
Arm/Group | 40 mg/m2 Prexasertib Exploratory Addendum
Number analyzed (Participants) | 15
nanograms per milliliter | 227 (68)

4. Secondary Outcome: Pharmacokinetics: Area Under the Concentration Curve of Prexasertib
Description: Pharmacokinetics: Area Under the Concentration Curve of Prexasertib
Time Frame: as for outcome 2
Population: All participants in Part A1 that received at least 1 dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg*h/mL
Groups:
- Cohort 1 Prexasertib (Platinum Sensitive Disease): Intravenous (IV) prexasertib (LY2606368) administered on day 1 of every 14 day cycle
- Cohort 2 Prexasertib (Platinum Resistant Disease): IV prexasertib (LY2606368) administered on day 1 of every 14 day cycle
- Cohort 3 Prexasertib Exploratory(Platinum Sensitive Disease): IV prexasertib (LY2606368) administered on Days 1, 2 and 3 of a 14-day cycle
Arm/Group | Cohort 1 Prexasertib (Platinum Sensitive Disease) | Cohort 2 Prexasertib (Platinum Resistant Disease) | Cohort 3 Prexasertib Exploratory(Platinum Sensitive Disease)
Number analyzed (Participants) | 56 | 60 | 15
mg*h/mL | 126 (154) | 1190 (95) | 1840 (35)

5. Secondary Outcome: Disease Control Rate: Percentage of Participants With a Best Overall Response of CR, PR, or Stable Disease (SD)
Description: Disease control rate (DCR) is defined as the percentage of participants achieving a best overall response of CR, PR, or SD as determined by RECIST 1.1. CR is defined as a disappearance of all target lesions and any pathological lymph nodes must have reduction in short axis to <10 mm and normalization of tumor marker results; PR is defined as at least a 30% decrease in the sum of diameter of target lesions, taking as reference the baseline sum diameters; SD is defined as neither sufficient shrinking to qualify as PR nor sufficient increase to qualify for PD.
Time Frame: Baseline through Disease Progression or Death from Any Cause to 28 months
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1 Prexasertib (Platinum Sensitive Disease) | Cohort 2 Prexasertib (Platinum Resistant Disease) | Cohort 3 Prexasertib Exploratory(Platinum Sensitive Disease)
Number analyzed (Participants) | 58 | 60 | 15
percentage of participants | 31 [12.6 to 31.4] | 20.0 [6.6 to 20.6] | 40.0 [10.2 to 48.4]

6. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS defined as the from randomization date to the first evidence of disease progression as defined by RECIST v1.1 or death from any cause. Progressive Disease (PD) was at least a 20% increase in the sum of the diameters of target lesions, with reference being the smallest sum on study and an absolute increase of at least 5 mm, or unequivocal progression of non-target lesions, or 1 or more new lesions. If a participant does not have a complete baseline disease assessment, then the PFS time was censored at the date of first dose, regardless of whether or not objectively determined disease progression or death has been observed for the participant. If a participant was not known to have died or have objective progression as of the data inclusion cutoff date for the analysis, the PFS time was censored at the last adequate tumor assessment date.
Time Frame: Baseline to Disease Progression or Death (up to 9 months)
Population: All randomized participants. 4 participants were censored from Prexasertib Cohort 1 and 1 participant from Prexasertib Cohort 3.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Prexasertib (Platinum Sensitive Disease) | Prexasertib (Platinum Resistant Disease) | Prexasertib Exploratory Addendum (Platinum Sensitive Disease)
Number analyzed (Participants) | 58 | 60 | 15
months | 1.41 [1.31 to 1.64] | 1.36 [1.25 to 1.45] | 1.58 [1.38 to 3.12]

7. Secondary Outcome: Duration of Response (DoR)
Description: DoR the time from the date of an objective response until Progressive Disease (PD): was at least a 20% increase in the sum of the diameters of target lesions, with reference being the smallest sum on study and an absolute increase of at least 5 mm, or unequivocal progression of non-target lesions, or 1 or more new lesions.
Time Frame: Date of CR or PR to Date of Disease Progression or Death Due to Any Cause up to 9 months
Population: Analysis was not performed due to only 3 responders in Cohort 1, no in Cohort 2 or 3. Individual data for Cohort 1 is presented.
Measure: Number; unit: days
Arm/Group | Cohort 1 Prexasertib (Platinum Sensitive Disease) | Cohort 2 Prexasertib (Platinum Resistant Disease) | Cohort 3 Prexasertib Exploratory(Platinum Sensitive Disease)
Number analyzed (Participants) | 58 | 60 | 15
days | NA — Individual DoR is 127, 172 and 153 days for 3 responders | NA — No responders | NA — No responders

8. Secondary Outcome: Overall Survival (OS)
Description: OS defined as from randomization date to the date of death due to any cause. For each participant who is not known to have died as of the data-inclusion cutoff date for overall survival analysis, OS time was censored on the last date the participant is known to be alive.
Time Frame: Baseline up to 28 months
Population: All randomized participants. 8 participants were censored from Cohort 1, 5 participants were censored from Cohort 2 and 4 participants censored from Cohort 3.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1 Prexasertib (Platinum Sensitive Disease) | Cohort 2 Prexasertib (Platinum Resistant Disease) | Cohort 3 Prexasertib Exploratory(Platinum Sensitive Disease)
Number analyzed (Participants) | 58 | 60 | 15
months | 5.42 [3.75 to 8.51] | 3.15 [2.27 to 5.52] | 7.26 [2.00 to 9.49]

9. Secondary Outcome: Change From Baseline in Lung Cancer Symptom Scale Score (LCSS)
Description: LCSS is a 9-item questionnaire, six measuring major symptoms for lung malignancies (appetite, fatigue, cough, dyspnea, hemoptysis and pain), and 3 summation items related to total symptomatic distress, activity status and overall quality of life. Participant responses were measured using visual analogue scales (VAS) with 100-mm lines. The LCSS total score was defined as the mean of the 9 items of the scale, each scored between 0 (for best outcome) to 100 (for worst outcome).
Time Frame: Baseline up to 9 months
Population: All participants in Cohort 1 and Cohort 2. Cohort 3 was added by protocol addendum and data were not collected with non missing baseline and post baseline scores.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cohort 1 Prexasertib (Platinum Sensitive Disease) | Cohort 2 Prexasertib (Platinum Resistant Disease)
Number analyzed (Participants) | 58 | 60
units on a scale | -2.8 (12.3) | -4.0 (10.2)

10. Secondary Outcome: Change From Baseline on the Average Symptom Burden Index (ASBI)
Description: ABSI was the mean score for the six major lung cancer symptoms (appetite, fatigue, cough, dyspnea, hemoptysis and pain), each scored between 0 (for best outcome) to 100 (for worst outcome).
Time Frame: Baseline up to 9 months
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cohort 1 Prexasertib (Platinum Sensitive Disease) | Cohort 2 Prexasertib (Platinum Resistant Disease)
Number analyzed (Participants) | 58 | 60
units on a scale | -3.0 (11.9) | -4.4 (11.1)

ADVERSE EVENTS:
Time Frame: up to 28 months
Description: All randomized participants who received at least 1 dose of study drug.
Groups:
- 40 mg/m2 Prexasertib Exploratory Addendum: IV 40 mg/m2 prexasertib (LY2606368) IV administered on Days 1, 2 and 3 of a 14-day cycle
Arm/Group | 105 mg/m^2 Prexasertib (Platinum Sensitive Disease) | 105 mg/m^2 Prexasertib (Platinum Resistant Disease) | 40 mg/m2 Prexasertib Exploratory Addendum
All-Cause Mortality (participants affected / at risk) | 10/56 | 7/60 | 11/15
Serious Adverse Events (participants affected / at risk) | 21/56 | 16/60 | 6/15
Other Adverse Events (participants affected / at risk) | 56/56 | 59/60 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 105 mg/m^2 Prexasertib (Platinum Sensitive Disease) (N=56) | 105 mg/m^2 Prexasertib (Platinum Resistant Disease) (N=60) | 40 mg/m2 Prexasertib Exploratory Addendum (N=15)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 8 (9) | 1 (1) | 2 (3)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (2) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 1 (2) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 2 (2) | 1 (1) | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Escherichia bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Parainfluenzae virus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 5 (9) | 0 (0) | 2 (3)
Pneumonia haemophilus (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 3 (3) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram qt prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 4 (7) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Cauda equina syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (2) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 105 mg/m^2 Prexasertib (Platinum Sensitive Disease) (N=56) | 105 mg/m^2 Prexasertib (Platinum Resistant Disease) (N=60) | 40 mg/m2 Prexasertib Exploratory Addendum (N=15)
Anaemia (Blood and lymphatic system disorders) | 28 (46) | 20 (36) | 9 (30)
Febrile neutropenia (Blood and lymphatic system disorders) | 5 (5) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 3 (4) | 6 (11) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 18 (30) | 18 (39) | 4 (11)
Thrombocytopenia (Blood and lymphatic system disorders) | 13 (27) | 9 (27) | 4 (11)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Eye haematoma (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 7 (9) | 6 (6) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 10 (14) | 5 (12) | 3 (3)
Nausea (Gastrointestinal disorders) | 15 (17) | 12 (16) | 3 (3)
Stomatitis (Gastrointestinal disorders) | 3 (4) | 2 (2) | 3 (3)
Vomiting (Gastrointestinal disorders) | 8 (11) | 7 (11) | 3 (3)
Asthenia (General disorders) | 8 (9) | 5 (7) | 2 (9)
Catheter site pain (General disorders) | 1 (1) | 0 (0) | 1 (1)
Fatigue (General disorders) | 16 (25) | 18 (25) | 6 (8)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 2 (2)
Non-cardiac chest pain (General disorders) | 7 (8) | 5 (5) | 0 (0)
Oedema peripheral (General disorders) | 4 (5) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 4 (4) | 5 (7) | 3 (3)
Oral candidiasis (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (3) | 2 (2) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (3) | 4 (8) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 5 (5) | 2 (2)
Blood cholesterol increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 1 (4) | 4 (5) | 0 (0)
Blood uric acid increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram qt prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 2 (5) | 5 (6) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 7 (18) | 6 (16) | 3 (5)
Neutrophil count decreased (Investigations) | 23 (62) | 26 (68) | 7 (38)
Platelet count decreased (Investigations) | 18 (49) | 23 (44) | 9 (36)
Weight decreased (Investigations) | 5 (5) | 3 (6) | 1 (1)
White blood cell count decreased (Investigations) | 14 (34) | 18 (59) | 5 (9)
Decreased appetite (Metabolism and nutrition disorders) | 13 (18) | 14 (20) | 6 (7)
Dehydration (Metabolism and nutrition disorders) | 6 (7) | 2 (3) | 1 (2)
Hyperuricaemia (Metabolism and nutrition disorders) | 3 (4) | 2 (3) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (4) | 3 (7) | 2 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 4 (5) | 2 (2) | 1 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 2 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 5 (6) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (5) | 1 (2) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (4) | 4 (5) | 0 (0)
Dizziness (Nervous system disorders) | 3 (5) | 1 (1) | 2 (2)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 5 (6) | 1 (2)
Confusional state (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (3) | 3 (3) | 1 (1)
Bronchial haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 16 (21) | 9 (9) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 (13) | 13 (14) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2016-03-15): https://cdn.clinicaltrials.gov/large-docs/80/NCT02735980/Prot_000.pdf
  • Statistical Analysis Plan (2016-05-16): https://cdn.clinicaltrials.gov/large-docs/80/NCT02735980/SAP_001.pdf